CLINICAL TRIAL: NCT00471900
Title: Physiolocal Effects of 6 Months DHEA Substitutional Therapy in Female Adrenal Failure in a Randomised, Placebo Controlled and Overcrossed Study.
Brief Title: Six Months DHEA Treatment in Female Adrenal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200110130
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dehydroepiandrosterone (DHEA)

SUMMARY:
DHEA is an adrenal deriven androgen precourser. The impact of DHEA substitution therapy in adrenal failure is unknown as well as the physiologically effects of DHEA is unknown. Effects of physiologically DHEA substitution is investigated in the model of female adrenal failure.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Adrenal insuficiency,
* Stable and safe anticonception,
* Stable hydrocortison substituation treatment.

Exclusion Criteria:

* Neoplastic and thromboembolic disease,
* Diabetes mellitus.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2001-10; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Quality of life parameteres, cardiovascular parameters, bodycomposition, exercise parameters, hormonal and serological parameters, fuel metabolisme. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christiansen, Professor, Study Director — Medical Dept. M, Aarhus University Hospital